CLINICAL TRIAL: NCT04539665
Title: Extended Mesenteric Excision in Ileocolic Resections for Crohn's Disease: A Multicenter Prospective Cohort Study
Brief Title: Extended Mesenteric Excision in Ileocolic Resections for Crohn's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Montreal General Hospital (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Sender Liberman MD, Dr. Sender Liberman, Associate Professor of Surgery and Oncology (McGill University), PI, Montreal General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: crohn's mesentery
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Crohn Disease; Recurrence; Crohn's Ileocolitis
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Prospective study arm involving an extended mesenteric ileocolic excision.
  Interventions: Procedure: Extended mesenteric resection.
- Control Arm (No Intervention): Historical controls from a retrospective chart review of patients who had a limited ileocolic resection.

INTERVENTIONS:
Procedure: Extended mesenteric resection. — Patients will undergo an ileocolic resection involving high ligation of the ileocolic pedicle, complete mobilization of the mesentery off of the retroperitoneum, and resection of the entire mesentery related to the specimen.
  Arms: Intervention Arm

SUMMARY:
The study is looking at the role of the mesentery in disease recurrence for ileocolic Crohn's disease. It is a prospective study that has been designed to perform extended mesenteric excision on patients undergoing their first ileocolic resection for Crohn's disease. Endoscopic recurrence will be monitored with the hypothesis that patients receiving extended mesenteric ileocolic resection will have reduced endoscopic recurrence at 6 months after resection.

DETAILED DESCRIPTION:
The current standard of care for ileocolic Crohn's disease (CD) is a limited mesenteric resection. There is growing, but still limited, evidence that extended mesenteric excision during ileocolic resection is beneficial in decreasing disease recurrence. We propose a prospective multicenter cohort study to better understand the role of extended mesenteric excision in ileocolic CD and how it affects disease recurrence. The primary outcome of this study will be the rate of endoscopic recurrence at 6 months in patients undergoing first-time resection for ileocolic CD. Secondary outcomes will include endoscopic recurrence at 18 months and rates of recurrence requiring surgery by 2 years. These outcomes will be compared to historical controls (limited mesenteric resection). Our hypothesis is that patients receiving extended mesenteric ileocolic resection will have reduced endoscopic recurrence at 6 months after resection. As seen in previous studies, advanced mesenteric and mucosal disease predicts increased surgical recurrence.

ELIGIBILITY:
Inclusion Criteria:

* adults >18 years old
* diagnosis of CD limited to the distal ileum/ileocolic region
* no previous ileocolic resection
* all forms of CD presentation will be included - stricturing, fistulizing, perforating etc.

Exclusion Criteria:

* previous ileocolic resection
* other sites of CD
* intraabdominal sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with endoscopic recurrence at 6 months | 6 months
  Endoscopic recurrence after extended mesenteric ileocolic resection

SECONDARY OUTCOMES:
Number of participants with endoscopic recurrence at 18 months | 18 months
  Endoscopic recurrence after extended mesenteric ileocolic resection.
Rates of recurrence requiring surgery by 2 years | 24 months
  Surgical recurrence after extended mesenteric ileocolic resection.
Rates of post-operative complications compared between study groups | 30 days
  Post-operative complications including: wound infections, anastomotic leak, intra-abdominal abscess, venous-thromboembolic complications, and primary ileus within 30 days of the first resection.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec